CLINICAL TRIAL: NCT03588598
Title: A Phase I Dose Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of SHC014748M in Patients With Relapsed or Refractory Indolent B-Cell Hematologic Malignancies.
Brief Title: Safety, Tolerability, and Pharmacokinetics of SHC014748M in Patients With Indolent B-Cell Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC014-I-01
Record Dates: First submitted 2018-06-28; First posted 2018-07-17 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); B-Cell Non-Hodgkin Lymphomas(NHL)
Keywords: CLL; SLL; NHL; SHC014748M; Phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHC014748M treatment (Experimental): SHC014748M capsule， 50, 100, 150, 200, 250 mg, QD, 28 days for each cycle
  Interventions: Drug: SHC014748M

INTERVENTIONS:
Drug: SHC014748M — a selective PI3Kδ inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of SHC014748M in patients with relapsed or refractory indolent B-cell hematologic malignancies.

DETAILED DESCRIPTION:
This is a phase I, sequential dose escalation followed by cohort expansion study of SHC014748M, an oral inhibitor of PI3K delta, in patients with relapsed or refractory indolent B-cell hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1.18- 75 years of age.

2.Histologically or cytologically confirmed diagnosis of relapsed or refractory indolent B-cell hematologic malignancies, including but not limited to CLL / SLL, FL (grade 1, 2 or 3a), or MZL.

3.Patients have received at least 1 prior regimen (at least 2 cycles).

4.Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.

5.Life expectancy ≥ 3 months.

6.Patients have at least 1 measurable lesion that measures ≥1.5 cm in a single dimension as assessed by CT or MRI.

7.Adequate organ function, as defined by the following values: ANC≥1.0×10^9/L； PLT≥50×10^9/L； Hb≥80 g/L； TBIL≤1.5×ULN； ALT and AST≤2.5×ULN； BUN and Cr≤1.5×ULN； LVEF≥50%； QTcF <450 ms for male, QTcF <470 ms for female；

8.Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose, and female subjects of childbearing potential have a negative pregnancy test at baseline.

9.Subjects did not participate in other clinical trials within 3 months prior to study entry.

Exclusion Criteria:

1. Disease progression after previous treatment with any PI3Kδ inhibitors.
2. Had any other anti-tumor treatment within 4 weeks prior to screening (including radiotherapy, chemotherapy, hormone therapy, surgery or targeted therapy).
3. Evidence of central nervous system involvement of the malignancy.
4. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, uncontrolled pleural effusion and ascites, uncontrolled diabetes, non-infectious pneumonia, and any other severe cardiovascular, respiratory, nervous and mental diseases.
5. Any of the severe heart diseases, including New York Heart Association (NYHA) Class II or greater heart failure, arrhythmias requiring medical treatment, and history of myocardial infarction or unstable angina within 6 months prior to screening.
6. Require any concomitant medication known to prolong the QT interval during the study.
7. Evidence of active bacterial, fungal, or viral infection.
8. Active infection with hepatitis B virus (HBV) (HBsAg positive, or HBsAg negative and HBV-DNA positive), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
9. Use of high-dose glucocorticoids (eg, ≥20 mg/day prednisone) or other immunosuppressants within 4 weeks prior to study entry.
10. Concomitant use of any strong inhibitors or inducers of CYP3A4.
11. Use of G-CSF or blood transfusion within 7 days before the hematology test at screening.
12. Prior autologous hematopoietic stem cell transplantation within 6 months prior to treatment initiation.
13. History of prior allogeneic hematopoietic stem cell transplantation.
14. Major surgery within 4 weeks prior to treatment initiation.
15. History of a non-lymphoma malignancy in the past five years except for the following: adequately treated cervical carcinoma in situ, local basal cell or squamous cell carcinoma of the skin.
16. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the drug or previous significant bowel resection that would preclude adequate absorption of the study drug.
17. History of hypersensitivity to drugs similar to the study drug or inactive excipients of the study drug.
18. Women who are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 1 month
Time to Peak Plasma Concentration（Tmax） | 1 month
Peak Plasma Concentration (Cmax) | 1 month
Half-life Time(t1/2) | 1 month
Area Under the Plasma Concentration Versus Time Curve (AUC) | 1 month

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months
Lymph Node Response (LNR) | up to 12 months
Time to Response (TTR) | up to 12 months
Progression-Free Survival (PFS) | up to 12 months
Duration of Response (DOR) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jie Jin, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No